CLINICAL TRIAL: NCT01437410
Title: Endoscopic Ultrasound-guided Fine Needle Aspiration of Solid Masses: Histological and Immunohistochemical Evaluation
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-01-044
Record Dates: First submitted 2011-09-09; First posted 2011-09-20 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Pancreatic Mass; Peripancreatic Mass
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — cytopathologic result acquired by endoscopic ultrasound-guided fine needle aspiration (EUS-FNA).

GROUPS / COHORTS (1):
- EUS-FNA
  Interventions: Procedure: EUS-FNA

INTERVENTIONS:
Procedure: EUS-FNA — tissue samples were harvested from 116 patients undergoing EUS-FNA of solid masses for cytologic smear and histological analysis.

SUMMARY:
The aim of this retrospective single center study was to evaluate the clinical utility of histological and immunohistochemical analyses of specimens obtained by endoscopic ultrasound-guided fine needle aspiration (EUS-FNA).

ELIGIBILITY:
Inclusion Criteria:

* We retrospectively reviewed medical records of patients who underwent EUS-FNA to evaluate solid pancreatic or peripancreatic lesions from January 2009 to July 2010

Exclusion Criteria:

* Patients with unavailable data

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent EUS-FNA to evaluate solid pancreatic or peripancreatic lesions from January 2009 to July 2010 in Samsung Medical Center,
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
the diagnostic accuracy of cytology, histology, and combined analysis of specimens obtained by EUS-FNA for pancreatic or peripancreatic solid masses | at least 6 months after surgery or clinical follow up
  The first, pre-op checked each diagnostic accuracy of cytology, histology, and combined analysis by EUS-FNA. and then, finaly diagnosis following surgery or clinical follow up for at least 6 months was re-check with diagnosic accuracy of cytology, histology, and combined analysis pre-diagnosed by EUS-FNA

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea